CLINICAL TRIAL: NCT02105584
Title: Prospective, Non-randomized, Safety and Efficacy Study of a New Occluder Design for Minimally Invasive Closure of the Left Atrial Appendage in Patients With Atrial Fibrillation
Brief Title: Prospective, Non-randomized, Safety and Efficacy Study of a New Occluder Design for Minimally Invasive Closure of the Left Atrial Appendage (LAA) in Patients With Atrial Fibrillation
Acronym: OLAAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Occlutech International AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OCC201202; CIV-13-09-011614 (Other: EUDAMED)
Record Dates: First submitted 2014-03-27; First posted 2014-04-07 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- LAA closure device (Experimental): Implantation of LAA closure device
  Interventions: Device: Implantation of LAA closure device

INTERVENTIONS:
Device: Implantation of LAA closure device
  Other Names: Occlutech LAA occluder in different sizes

SUMMARY:
This is a prospective, non-randomized, study of the safety and efficacy of the Occlutech® LAA occluder indicated for percutaneous LAA closure in adult male or female patients with atrial fibrillation. Safety and efficacy will be assessed at day 1, 30 and 90, and after 1 year following implantation of an Occlutech® LAA Occluder.

ELIGIBILITY:
Inclusion Criteria:

* Documented paroxysmal, persistent or chronic non-valvular AF
* Calculated CHA2DS2 -VASC score equal or greater than 2 and/or HAS-BLED score equal or greater than 2
* Patients eligible or non-eligible for lifelong, oral anticoagulation therapy
* Life expectancy of at least 1 year
* Written, informed consent by the patient or her/his legally-authorized representative for participation in the study

Exclusion Criteria:

* Suspected or known intracardiac thrombus
* NYHA Class IV CHF
* Patients who has unstable and intractable angina pectoris
* ASD and/or atrial septal repair or closure device
* Recent myocardial infarction within 3 months
* Severe valvular heart disease, or implanted mechanical valve prosthesis
* Large PFO with significant atrial septal aneurysm
* Planned ablation procedure within 30 days of Occlutech LAA occluder® implant
* Resting heart rate > 110 bpm
* Allergy to Nitinol, which is a result of nickel and/or titanium allergies
* Stroke/TIA within the last 30 days
* Thrombocytopenia, thrombocytosis, leukopenia, or anemia
* Symptomatic carotid artery disease
* LVEF < 30%
* Mitral valve stenosis

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2014-04; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Successful implantation of the Occlutech LAA closure device with less than 7% occurrence of major complications. | 12 months
  A major complication is defined as an event that results in death, procedure related stroke, systemic embolism, device embolisation, pericardial effusion (cardiac tamponade), or other major bleeding requiring invasive treatment or blood transfusions.

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Brachmann, Prof, Principal Investigator — Klinikum Coburg
Locations (7):
- Germany (6):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Kardiologie Universitätsklinikum Bonn, Bonn
  - Medizinische Klinikum Coburg, Coburg
  - CardioVascular Center Frankfurt, Frankfurt
  - Klinik für Innere Medizin Kardiologie Herzzentrum Leipzig GmbH, Leipzig
  - University Medical Center of Johannes Gutenberg-University Mainz, Mainz
- NHS Trust (ICHNT) Hammersmith Hospital London, London, United Kingdom